CLINICAL TRIAL: NCT04671459
Title: A Phase II Trial of Tumor Treating Fields (TTFields) Concomitant With Radiosurgery for the Treatment of Recurrent, Bevacizumab-naïve Glioblastoma
Brief Title: TTFields and Radiosurgery of Recurrent Glioblastoma +/- 18F-Fluoro-Ethyl-Thyrosine
Acronym: TaRRGET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Franciszek Lukaszczyk Memorial Oncology Center (Other)
Collaborators: NovoCure GmbH (Industry)
Responsible Party: Principal Investigator, Maciej Harat, dr hab. n. med. Maciej Harat prof. UMK, Prof. Franciszek Lukaszczyk Memorial Oncology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB 2020
Record Dates: First submitted 2020-12-05; First posted 2020-12-17 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Glioblastoma Multiforme; Recurrent Glioblastoma
Keywords: Glioblastoma; SRS; GBM; recurrent GBM; recurrence; stereotactic radiosurgery; Radiosurgery; FET-PET; 18F-fluoro-etyl-thyrosine; TTFields; Optune
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Spermine Synthase; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase II trial enrolling participants with recurrences or progressive tumor, who will be treated with radiosurgery and TTFields. The investigators will attempt to enroll the maximum number of patients and expect to enroll 40 subjects. All subjects will receive TTFields and radiosurgery plus/minus FET PET imaging to define tumor volume.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TTFields and SRS based on MRI or FET-PET (Experimental): All subjects will receive TTFields and radiosurgery plus/minus FET PET imaging to define tumor volume.
  Interventions: Combination Product: TTFields and SRS

INTERVENTIONS:
Combination Product: TTFields and SRS — SRS procedure will be delivered within 7 days after start of TTFields therapy . A 5-day SRS regimen is allowed. TTFields should be interrupted in time of SRS and start immediately after.
  Other Names: Optune, Stereotactic Radiosurgery

SUMMARY:
All patients will receive TTFields therapy and additionally Stereotactic Radiosurgery . Radiosurgery will be based on MRI and FET-PET or MRI alone. Addition of FET-PET will be preferred option.

DETAILED DESCRIPTION:
Almost all GBM patients experience recurrent disease. Stereotactic radiosurgery (SRS),at recurrence, has limitations due to the invasive nature of glioblastoma. TTFields may decrease the tumor aggressiveness outside the target area potentially by multiple pathways, including immunogenic cell death and DNA repair inhibition sensitizing to radiation. We hypothesize that combined SRS and TTFields will be complementary, improving outcomes with minimal toxicity.

In this open-label, phase II trial 40 participants with recurrence will be treated with SRS and TTFields, starting in 2020. Recurrence will be defined on FET-PET or MRI using RANO criteria.

All patients will begin treatment within 14 days from baseline imaging evaluation and at maximum 42 days from screening.

The attempt to obtain the Methyl-guanine methyl-transferase (MGMT) gene promoter methylation and IDH1 and IDH2 mutation from primary tumor are made during the study whenever not defined before entering to the study.

TTFields treatment will be initiated as in clinical routine at patients home. Admission to hospital will not be necessary.

SRS must be delivered within 7 days of TTFields start. A 5-day SRS regimen is allowed. TTFields should be interrupted only during SRS. The sample size of the study was calculated for the comparison of survival against a historical control.Overall survival will be stratified by volume, PET-based treatment, SVZ invasion, MGMT methylation status, time to first progression, and TTFields compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's written informed consent (IC) obtained at the latest the day after planning MRI;
2. Legal capacity: patient can understand the nature, significance, and consequences of the study;
3. Age ≥18 years (no upper age limit);
4. Karnofsky Performance Score (KPS) ≥ 70;
5. Recurrence of GBM (WHO grade IV) based on RANO criteria or GBM after subtotal resection of recurrence with macroscopic residual tumor;
6. Histological confirmation of GBM at initial or secondary diagnosis;
7. Previous radiotherapy of glioma with a total dose of 59.4 - 60 Gy (single dose 1.8 - 2.0 Gy) and chemotherapy with temozolomide;
8. At least 6 months between the end of the first course of radiotherapy and radiosurgery;
9. Recurrent tumor visible on FET-PET and/or T1Gd-MRI, with the maximum diameter up to 5 cm by either technique (in case of multifocal tumors, the sum of all diameters must be 5 cm on FET-PET and T1Gd-MRI);
10. Start of TTFields before radiosurgery;
11. Disease free from other cancers for ≥ 5 years;
12. Adequate haematologic, renal and hepatic function (absolute neutrophil count ⩾1000/mm3; haemoglobin ⩾100 g/L platelet count, ⩾100,000/mm3; serum creatinine level ⩽1.7 mg/dL (<150 μmol/L); total serum bilirubin level ⩽ the upper limit of normal and liver-function values, <3 times the upper limit of normal);

Exclusion Criteria:

1. Recent (≤ 4 weeks before IC) histological result showing no tumor recurrence;
2. Previous treatment of GBM with bevacizumab;
3. Chemotherapy or molecular targeted therapies planned before diagnosis of further tumor progression after study intervention
4. Simultaneous participation in other interventional trials which could interfere with this trial and/or participation in a clinical trial within the last thirty days before the start of this study and/or previous participation (randomization) in this study;
5. Pregnancy, nursing, or patient not willing to prevent a pregnancy during treatment;
6. Known or persistent abuse of medication, drugs or alcohol;
7. Known allergy against the MRI contrast agent gadolinium or the PET tracer 18F-FET or against any of the components;
8. Evidence of increased intracranial pressure (midline shift >5 mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness);
9. Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
10. Gross total resection of recurrence confirmed with postoperative MRI and negative FET-PET result
11. Other malignancies ,except for non-melanomatous skin cancers, or carcinoma in-situ of uterus, cervix or bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-26 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
1-year survival rate | 12 Months
  Survival will be measured from date of enrollment until date of death

SECONDARY OUTCOMES:
Radiation necrosis range | 12 months
  The percentage of patients who had radiation necrosis
Progression free survival (PFS) | 12 moths
  PFS will be measured from the date of enrollment to date of progression (in months) based on RANO citeria.
Steroid needs until treatment failure | 12 months
  The analysis will be performed based on the steroid doses reported in time of enrollment to date of progression or one year after
Patterns of failure | 12 months
  The analysis will be performed based on location of failure in relation to target volume
Objective response rates | 12 months
  The percentage of patients who had either complete response or partial response per RANO criteria following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Harat, MD PhD, Principal Investigator — Prof. Franciszek Lukaszczyk Memorial Oncology Center
Locations (1):
- The Franciszek Lukaszczyk Oncology Center, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No
IPD and all supporting data will be available upon request.